CLINICAL TRIAL: NCT01067456
Title: Diagnostic Value of Comprehensive Cardiothoracic Dual Source CT for the Early Triage of Patients With Undifferentiated Acute Chest Pain
Brief Title: Comprehensive Cardiothoracic Dual Source CT for the Early Triage of Patients With Acute Chest Pain
Acronym: CAPTURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bracco Diagnostics, Inc (Industry)
Responsible Party: Principal Investigator, Udo Hoffmann, MD MPH, Director, Cardiac Imaging, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008P000389
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Chest Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized diagnostic trial, two arms
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dedicated CT arm (No Intervention): Subjects in this arm will continue to receive standard of care - that is the dedicated CT protocol to rule out either aortic dissection or acute coronary syndrome or pulmonary embolism.
- Comprehensive Cardiothoracic CT arm (Experimental): The intervention consisted in a change of the routine CT protocol (as in dedicated CT protocol) to a comprehensive cardiothoracic CT protocol which includes changes in contrast injection and coverage to enable evaluation of the presence of acute coronary syndrome/aortic dissection/pulmonary embolism in a single scan.
  Interventions: Radiation: Comprehensive Cardiothoracic CT arm

INTERVENTIONS:
Radiation: Comprehensive Cardiothoracic CT arm — Subjects in this arm will receive the comprehensive cardiothoracic CT to rule out aortic dissection/pulmonary embolism/acute coronary syndrome in a single scan.
  Arms: Comprehensive Cardiothoracic CT arm

SUMMARY:
The purpose of this research is to determine the efficiency of a single dual source computed tomography (CT-DSCT) protocol to establish or exclude acute coronary syndrome (ACS), pulmonary embolism (PE) or aortic dissection (AD) as compared to the individual protocols. Endpoints aim to compare the rate of emergency department (ED) discharge, length of hospital stay, the diagnostic imaging test utilization, and the costs between the comprehensive and the standard protocol strategy in patients with undifferentiated chest discomfort or shortness of breath with a component of chest discomfort.

DETAILED DESCRIPTION:
Undifferentiated chest pain is one of the most common complaints in the acute care setting, accounting for over five million emergency department (ED) visits in the U.S. each year. Moreover, early and accurate triage of these patients remains difficult as neither the chest pain history, a single set of biochemical markers for myocardial necrosis, or the initial 12-lead electrocardiogram (ECG), alone or in combination, identify a group of patients that can be safely discharged without further diagnostic testing. As a result, patients presenting to the ED with undifferentiated chest pain are often evaluated with multiple examinations to exclude the presence of myocardial infarction (MI),pulmonary embolism (PE), and/or aortic dissection (AD).

While contrast-enhanced spiral computed tomography angiography (CTA) has become a standard procedure in the evaluation of the presence of PE and AD, it was only within the past few years that noninvasive detection of coronary artery stenosis with CTA has become feasible. Coronary CTA has been proven to be an effective tool to rule out CAD with reported sensitivities of 93-99% and specificities of 95-97% as compared to invasive coronary angiography.

Recent data from our Rule Out Myocardial Infarction by Computer Assisted Tomography (ROMICAT) study indicates that coronary CTA accurately rules out acute coronary syndrome (ACS) in patients with acute chest pain and therefore may enhance the diagnostic work up of chest pain patients in the ED. Moreover, this study demonstrated the distribution of several CT-angiographic patterns of CAD which may change management of subjects with inconclusive initial ED evaluation admitted to the hospital. For example, CTA demonstrated the absence of any CAD in 50% of the patients. None of the subjects without any CAD on CTA developed unstable angina or had an MI during index hospitalization. Furthermore, none of these patients had any MACE over the next six months, confirming previous observations in ACS patients. These data suggest that 50% of hospital admissions could be saved. Another recent study our group has demonstrated that an individually tailored ECG-gated CT protocol with a single contrast injection permits simultaneous visualization of the coronary arteries, thoracic aorta, and pulmonary arteries with excellent image quality.

The very recent introduction of dual source CT (DSCT) technology offers a two-fold improvement in temporal resolution as compared to the standard 64-slice CTA that was used for these studies (83ms vs. 165ms, respectively). This significant improvement in temporal resolution allows for the acquisition of diagnostic images with higher and irregular heart rates, precluding the need for intravenous beta blockade. Given the improved temporal resolution and faster acquisition time, the amount of radiation exposure can be markedly reduced in many patients.

With the need to improve triage of patients with undifferentiated chest pain and the advantages offered by DSCT technology, several observational case series have suggested the feasibility of a comprehensive thoracic DSCT (CT-DSCT) to simultaneously evaluate the coronary arteries, thoracic aorta, and pulmonary arteries. Whether this will result in an improvement of patient management and test utilization remains unclear as compared to a standard ED evaluation protocol needs to be evaluated.

Thus, the purpose of this research is to determine the efficiency of a single CT-DSCT protocol to establish or exclude MI, PE, or AD as compared to the individual protocols. Endpoints aim to compare the rate of ED discharge, length of hospital stay, the diagnostic imaging test utilization, and the costs between the comprehensive and the standard protocol strategy in patients with undifferentiated chest discomfort or shortness of breath with a component of chest discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Males or females >30 years of age in sinus rhythm
* Willing and able to provide written informed consent
* Undifferentiated chest discomfort or shortness of breath with a component of chest discomfort within the last 24 hours
* Intermediate likelihood of MI, pulmonary embolism (PE), or aortic dissection (AD) as determined by ED providers after completion of standard initial clinical evaluation
* ED providers independently decide that the patient's care plan should include a coronary, PE, or AD CT.
* Female patients must be either of non-childbearing potential (i.e., surgically sterilized or post menopausal [≥ 12 consecutive months without menses]) or must have a negative pregnancy test

Exclusion Criteria:

* Positive cardiac biomarkers (elevated serum creatine phosphate (CK) with elevated CK-MB isoform and/or elevated troponin)
* Diagnostic ECG changes (e.g., >1 mm ST-segment elevation or depression in two anatomically contiguous leads)
* Known history of CAD (i.e., past myocardial infarction, prior coronary stent Placement, and/or coronary artery bypass graft surgery)
* Known history of thoracic aortic disease (i.e., thoracic aortic aneurysm > 5cm in diameter, history of aortic dissection, and/or history of thoracic aortic aneurysm repair (via open surgery or stent-graft placement))
* Known history of pulmonary embolism
* Heart rate > 100 beats per minute
* Systolic blood pressure <105 mmHg
* Oxygen saturation < 90%
* Any cardiac arrhythmia causing hemodynamic compromise
* Serum creatinine clearance <60 mL/min by Cockcroft-Gault
* Known allergy to iodinated contrast agents
* Subjects on metformin therapy that are unable or unwilling to discontinue therapy for 48 hours after CT procedure

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Hoffmann, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Emergency Department, 9-month enrollment period starting January 2008
Groups:
- Comprehensive Cardiothoracic CT Arm: Subjects in this arm receive a comprehensive cardiothoracic CT to evaluate the presence of acute coronary syndrome/aortic dissection/pulmonary embolism in a single scan.
Period: Overall Study
Arm/Group | Dedicated CT Arm | Comprehensive Cardiothoracic CT Arm
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Comprehensive Cardiothoracic CT Arm: Subjects in this arm receive a comprehensive cardiothoracic CT to evaluate the presence of acute coronary syndrome/aortic dissection/pulmonary embolism in a single scan.
  Comprehensive Cardiothoracic Dual Source CT (DSCT) arm: Subjects in this arm will receive the comprehensive cardiothoracic DSCT to rule out aortic dissection/pulmonary embolism/acute coronary syndrome in a single scan.
- Total: Total of all reporting groups
Arm/Group | Dedicated CT Arm | Comprehensive Cardiothoracic CT Arm | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 53 (11) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 20 | 23 | 43
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Time Frame: Index Hospitalization (within 48 hours)
Measure: Median (Inter-Quartile Range); unit: Hours
Groups:
- Comprehensive Cardiothoracic CT Arm: Subjects in this arm receive a comprehensive cardiothoracic CT to evaluate the presence of acute coronary syndrome/aortic dissection/pulmonary embolism in a single scan.
  Comprehensive Cardiothoracic DSCT arm: Subjects in this arm will receive the comprehensive cardiothoracic DSCT to rule out aortic dissection/pulmonary embolism/acute coronary syndrome in a single scan.
Arm/Group | Dedicated CT Arm | Comprehensive Cardiothoracic CT Arm
Number analyzed (Participants) | 30 | 29
Hours | 7.63 [5.38 to 28.23] | 8.20 [5.32 to 30.08]
Statistical Analysis 1: Comparison: Dedicated CT Arm vs Comprehensive Cardiothoracic CT Arm; Test type: Superiority or Other; p = 0.79, t-test, 2 sided; Median Difference (Final Values) = 0.57

2. Secondary Outcome: Direct Hospital Discharge Without Imaging
Description: Number of patients discharged without imaging
Time Frame: Index Hospitalization (within 48 hours)
Measure: Count of Participants; unit: Participants
Groups:
- Dedicated CT Arm: Standard CT either cardiac, PE or aortic dissection CT
- Comprehensive Cardiothoracic CT Arm: That is the interventional arm with the new protocol
Arm/Group | Dedicated CT Arm | Comprehensive Cardiothoracic CT Arm
Number analyzed (Participants) | 30 | 29
Participants | 21 | 20

3. Secondary Outcome: Cost of Care
Description: Cost of stay in USD
Time Frame: Index Hospitalization (within 48 hours)
Measure: Median (Inter-Quartile Range); unit: cost in USD
Arm/Group | Dedicated CT Arm | Comprehensive Cardiothoracic CT Arm
Number analyzed (Participants) | 30 | 29
cost in USD | 1724 [1277 to 4208] | 1898 [1554 to 5116]

ADVERSE EVENTS:
Groups:
- Dedicated CT Arm: Subjects in this arm continued to receive standard of care - that is the dedicated CT protocol to rule out either aortic dissection or acute coronary syndrome or pulmonary embolism.
- Comprehensive Cardiothoracic CT Arm: Subjects in this arm received a comprehensive cardiothoracic CT to evaluate the presence of acute coronary syndrome/aortic dissection/pulmonary embolism in a single scan.
Arm/Group | Dedicated CT Arm | Comprehensive Cardiothoracic CT Arm
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dedicated CT Arm (N=30) | Comprehensive Cardiothoracic CT Arm (N=29)
Myocardial Infarction (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No